CLINICAL TRIAL: NCT07153380
Title: Critical Assessment of Respiratory, Physical and Emotional Distress in Critically Ill Patients With and Without Invasive Mechanical Ventilation
Brief Title: Evolution of Physical and Emotional Distress in ICU
Acronym: CARE-ICU
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Elisabet Doña-López, Researcher, Corporacion Parc Tauli
Other Study IDs: 2025/5057
Record Dates: First submitted 2025-07-29; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: ICU Ill Patients; Critical Illness
Keywords: ICU patients; dypnea; emotional state ICU; pain; ICU physical distress; ICU emotional distress; ICU admission
MeSH Terms: conditions — Critical Illness; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CARE-ICU: Critically ill patients during ICU admission

SUMMARY:
Emotional distress is prevalent in ICU patients and may be influenced by physical symptoms such as dyspnea and pain, yet its evolution and interactions during ICU stay remain insufficiently explored. The main objective of this study is to investigate the trajectory of anxiety, sadness, dyspnea, and pain during ICU stay, as well as their associations with clinical and demographic factors. Moreover, the investigators will study the impact of emotional distress during ICU admission in the cognitive status of the ICU survivors at discharge.

In this study the investigators will recover the data of 62 ICU patients who participated in 3 different studies lead by the research line of Characterization and Managment of the Post-Intensive Care Syndrome from the I3PT research Group of Translational Research in the Physiopathology of the Critically Ill Patients. In the 3 studies, emotional distress (anxiety and sadness), dyspnea, and pain were evaluated daily using visual analog scales once adequate consciousness was achieved (RASS -1 to +1). Cognitive status at ICU discharge was assessed using the Montreal Cognitive Assessment (MoCA). The datasets of the 3 studies will be revised and a new database will be generated with participants who have an assessment of emotional distress for at least 80% of the ICU length of stay with an optimal level of consciousness (RASS >-1). New mixed-effects models will be used to explore the evolution of emotional and physical distress during ICU admission and the associations with invasive mechanical ventilation (IMV), and other demographic and clinical variables. Expected results: the investigators expect a better understanding of the evolution of anxiety and sadness symptoms during ICU stay and its relationship with the level of dyspnea and pain experienced by the critically ill patients during admission.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Admitted to the ICU for at least ≥ 24 hours

Exclusion Criteria:

* Previous cognitive impairment or dementia
* Prior history of neurological disease (including brain damage at admission)
* Severe psychiatric disorder (including substance use disorder)
* Intellectual disability
* Non-Spanish speaker
* Life expentancy <12 months
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients admitted to Parc Taulí Hospital
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Emotional distress | During ICU admission
  Daily levels of anxiety and depression symptoms- Assessed by Visual Analog Scale (VAS).
  The assessment is carried out once the admitted critically ill patient reaches a minimum level of consciousness (Richmond Agitation Sedation Scale ≥-1).
Physical distress | During ICU admission
  Daily levels of dyspnea and pain. - Assessed by Visual Analog Scale (VAS). The assessment is carried out once the admitted critically ill patient reaches a minimum level of consciousness (Richmond Agitation Sedation Scale ≥-1).

SECONDARY OUTCOMES:
Cognitive status | From the first documented data on discharge from the ICU for the first subject included in the study, to the last documented data on discharge from the ICU for the last patient included in the study, evaluated up to 24 months.
  MoCA test

CONTACTS AND LOCATIONS:
Locations (1):
- I3PT Instituto de Investigación e Innovación Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dona-Lopez E, Godoy-Gonzalez M, Navarra-Ventura G, Fernandez-Olivares A, Goma G, Estela Esteve J, De Haro C, Diaz Santos E, Salarbous L, Jodar M, Blanch L, Lopez-Aguilar J, Fernandez-Gonzalo S. Trajectories of emotional and physical distress during ICU stay and their association with clinical factors and cognitive status at discharge. Sci Rep. 2026 Jan 27. doi: 10.1038/s41598-026-36684-y. Online ahead of print. PMID 41588070